CLINICAL TRIAL: NCT02816775
Title: Hemodynamic Responses to Tracheal Intubation Direct Laryngoscope and Videolaryngoscope in Elderly Patients: A Randomized, Controlled Trial
Brief Title: Hemodynamic Responses to Tracheal Intubation Direct Laryngoscope and Videolaryngoscope in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ülkü Özgül, Associate professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Ulku2
Record Dates: First submitted 2016-06-20; First posted 2016-06-29 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Aged Patients
Keywords: hemodynamics; QT interval

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Laryngoscope (Active Comparator): Group Laryngoscope; intubation will be made by Macintosh laryngoscope
  Interventions: Device: Macintosh Laryngoscope
- Group Videolaryngoscope (Active Comparator): Group Videolaryngoscope; intubation will be made by McGRATH Videolaryngoscope
  Interventions: Device: McGRATH Videolaryngoscope

INTERVENTIONS:
Device: Macintosh Laryngoscope — After induction of anesthesia, tracheal intubation will made by Macintosh Laryngoscope
  Arms: Group Laryngoscope
Device: McGRATH Videolaryngoscope — After induction of anesthesia, tracheal intubation will made by McGRATH Videolaryngoscope
  Arms: Group Videolaryngoscope

SUMMARY:
The intubation response to airway manipulation during direct laryngoscopy can cause hypertension, dysrhythmias and increased intracranial and intraocular pressures. This intense physiological response is proven to be associated with adverse outcomes especially in elderly patients. Increased QT dispersion is associated with increased risk of ventricular arrhythmias, which may increase the risk of sudden death caused by life-threatening arrhythmias. McGrath Videolaryngoscope would generate a lesser haemodynamic response than the conventional method of direct laryngoscopy. The objective of this study was to compare the hemodynamic response and QT during following tracheal intubation, using videolaryngoscope or direct laryngoscope to intubation. The postoperative airway morbidities is the investigators secondary outcome.

DETAILED DESCRIPTION:
Ninety patients, aged over 65 years, scheduled for elective surgery under general anesthesia requiring tracheal induction will be included in this study.

All patients will divided into two groups by a sealed envelope technique, Group Laryngoscope; n = 45 and Group Videolaryngoscope; n = 45 to receive tracheal intubation using either a Macintosh laryngoscope (Group L) or a McGRATH videolaryngoscope (Group V).

Hemodynamic data will evaluated by an anesthesiologist who was blinded to the study group affiliations. Evaluation of ECG will performed by a cardiologist.

None of the patients will premedicated with any drug. Standard monitors, including ECG (lead II), noninvasive systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP) and peripheral oxygen saturation (SpO2) measurements will be and mallampati classification, thyromental distance and mouth opening will be evaluated. After preoxygenation, anesthesia will induced with propofol 1.5 mg/kg. After loss of consciousness, rocuronium 0.5 mg/kg will injected intravenously (IV). Two minutes after rocuronium administration, fentanyl 2.0 μg/kg was given to each patient, and intubation will attempted with the direct laryngoscopy or McGrath Videolaryngoscopy. Anesthesia will maintained with sevoflurane in a mixture of 50% oxygen in 50% nitrous oxide.

The following parameters will measured by a blind observer: number of intubation trials, intubation time (from insertion of the intubation device into the mouth to capnographic confirmation), airway trauma (detection of blood drops in the mouth, lip or the tube after removal). SBP, DBP, MAP heart rate and electrocardiography (ECG) will recorded at the following time points: before induction of anesthesia (pre-induction, T0), before tracheal intubation (post-induction, T1), 1,3,5 min post-intubation (T2, T3, T4, respectively).

A 12-lead surface ECG was obtained from each subject while placed in the supine position. The 12-lead ECG was recorded at a standardized article speed of 50 mm/sec and 2.0 millivolt/cm. Measurement of QT interval duration will carried out manually using a caliper.

Pharyngolaryngeal injury in all patients will assessed by asking about sore throat and hoarseness 24 h after the surgery using an 4-point scale: none, mild, moderate and severe.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective surgery under general anesthesia requiring tracheal intubation

Exclusion Criteria:

* hypertension,
* cardiopulmonary disease,
* diabetes mellitus,
* a predicted problematic airway,
* morbid obesity,
* the use of medications known to affect blood pressure and heart rate as β-adrenergic blockers

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
mean blood pressure | Change from baseline mean blood pressure at 30 minutes
  The patient's blood pressure should be measured and recorded at 5-minute intervals during the first 30 minutes of the operation.

SECONDARY OUTCOMES:
QT interval | Change from baseline QT interval at 30 minutes
  The QT interval in the ECG recordings in the first 30 minutes will be evaluated.
heart rate | Change from baseline heart rate at 30 minutes
  The patient's heart rate should be measured and recorded at 5-minute intervals during the first 30 minutes of the operation.
Number of participants with treatment-related adverse events as assessed by 4- point scale | From extubation until postoperative 24 hours
  Sore throat and hoarseness is graded as: none, mild, moderate, severe

CONTACTS AND LOCATIONS:
Overall Officials: Türkan Toğal, Prof., Study Director — Inonu University Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tempe DK, Chaudhary K, Diwakar A, Datt V, Virmani S, Tomar AS, Mohandas A, Mohire VB. Comparison of hemodynamic responses to laryngoscopy and intubation with Truview PCD, McGrath(R) and Macintosh laryngoscope in patients undergoing coronary artery bypass grafting: A randomized prospective study. Ann Card Anaesth. 2016 Jan-Mar;19(1):68-75. doi: 10.4103/0971-9784.173023. PMID 26750677